CLINICAL TRIAL: NCT03399461
Title: Understanding of the Patient and Caregiver Experience of Wiskott-Aldrich Syndrome (WAS)
Brief Title: Targeted Literature Review and Subject Interviews in Wiskott-Aldrich Syndrome (WAS)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 208034
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Wiskott-Aldrich Syndrome
Keywords: United States; United Kingdom; Wiskott-Aldrich Syndrome; Caregiver; Interview; immune deficiency; France
MeSH Terms: conditions — Wiskott-Aldrich Syndrome; Immunologic Deficiency Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Approximately 8 subjects with WAS between ages of 12 to 30 years will be included in Group 1.
  Interventions: Other: Patient Interview guide; Other: Sociodemographic questionnaire; Other: Pediatric quality of life (PedsQL) questionnaire; Other: Clinical questionnaire
- Group 2: Approximately 8 primary caregivers of subjects with WAS between ages 8 to 30 years will be included in Group 2.
  Interventions: Other: Caregiver interview guide; Other: Sociodemographic questionnaire; Other: Pediatric quality of life (PedsQL) questionnaire; Other: Clinical questionnaire
- Group 3: Approximately 5 primary caregivers of subjects with WAS under the age of 8 years will be included in Group 3.
  Interventions: Other: Caregiver interview guide; Other: Sociodemographic questionnaire; Other: Pediatric quality of life (PedsQL) questionnaire; Other: Clinical questionnaire

INTERVENTIONS:
Other: Patient Interview guide — The interviewer will conduct the interview for subjects with WAS using a semi-structured patient interview guide.
  Groups: Group 1
Other: Caregiver interview guide — The interviewer will conduct the interview for caregivers of subjects with WAS using a semi-structured caregiver interview guide.
  Groups: Group 2; Group 3
Other: Sociodemographic questionnaire — At the end of interview, subjects will be required to complete subject or caregiver versions of country-specific sociodemographic questionnaire.
Other: Pediatric quality of life (PedsQL) questionnaire — The PedsQL is a validated generic measure of health-related quality of life (HRQOL) in children, adolescents, and young adults with acute and chronic health conditions. At the end of interview, subjects will be required to complete subject or caregiver versions of PedsQL questionnaire.
Other: Clinical questionnaire — At the end of interview, subjects will be required to complete subject or caregiver versions of clinical questionnaire.

SUMMARY:
WAS is a rare primary immune deficiency disease caused by genetic mutation and is more common in males than females. The purpose of this study is to understand experiences of WAS subjects and caregivers to identify important concepts of interest that could be measured in future Phase IIIb trials. This is a qualitative cross-sectional study that will include a sample of approximately, 8 subjects with WAS and 13 caregivers of subjects with a diagnosis of WAS in the United States, United Kingdom and France. A 60 to 90 minute open-ended interview will be conducted over the telephone or video conference that will be audio-recorded for subsequent transcription. The aim of these interviews is to obtain subject and caregiver perspectives on the impact of WAS and its associated treatments on quality of life and experiences of living with WAS.

ELIGIBILITY:
Inclusion Criteria:

Subjects:

* Male adolescents or young adults ranging in age from 12 through 30 years old.
* Diagnosis of WAS defined by WAS genetic mutation with a clinical score >=1 or self-reported disease severity.
* Subjects who are "conservatively managed" or have not received treatment for WAS; a maximum of 5 subjects who have received a hematopoietic stem cell transplant within the preceding two years.
* Able to read, speak, and understand English or French sufficiently to complete all assessments.
* Willing and able to participate in an audio-recorded, telephone or video conference session, including adherence to the interview instructions and completion of all questionnaires.
* Parent/guardian/patient signed informed consent.

Caregivers:

* Caregivers of children >=2 years of age diagnosed with WAS; at least 5 caregivers of subjects under the age of 8.
* Caregivers of subjects with a diagnosis of WAS defined by WAS genetic mutation with a clinical score >=1 or self-reported disease severity.
* Caregivers of subjects who are "conservatively managed" or have not received treatment for WAS; At least 2 caregivers of subjects who have received a hematopoietic stem cell transplant within the preceding two years.
* Caregivers are defined as primary caregiver.
* Able to read, speak, and understand English or French sufficiently to complete all assessments.
* Willing and able to participate in an audio-recorded, telephone or video conferencing interview session, including adherence to the interview instructions and completion of all questionnaires.
* Caregivers of Wiskott-Aldrich patients can be of any age or gender and do not have to follow the patient inclusion criteria, as long as their child/patient meets the inclusion criteria, as outlined.

Exclusion Criteria:

Subjects

* Subjects who have previously received gene therapy treatment Caregivers
* Caregivers of subjects who have previously received gene therapy treatment
* Professional caregivers (that is, at home nurse or equivalent).

Ages: 12 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: A convenience sample of approximately, 21 subjects with WAS and primary caregivers of WAS subjects will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Number of subject reported perspectives on WAS | Up to 90 minutes
  Open-ended interviews will be conducted in adolescent and adult subjects to understand their perspective on WAS.
Number of caregiver reported perspectives on WAS | Up to 90 minutes
  Open-ended interviews will be conducted in caregivers of subjects with WAS to understand their perspective on WAS.
Number of subject reported preventative measures taken to avoid infection and bleeding | Up to 90 minutes
  The preventative measures taken to avoid infection and bleeding as reported by subjects during open-ended interviews will be summarized.
Number of caregiver reported preventative measures taken to avoid infection and bleeding | Up to 90 minutes
  The preventative measures taken to avoid infection and bleeding as reported by caregivers during open-ended interviews will be summarized.
Number of subject reported awareness on the risk of disease | Up to 90 minutes
  Open-ended interviews will be conducted in adolescent and adult subjects to understand their awareness on the risk of disease (that is, risk of future complications and potential rapid decline).
Number of caregiver reported awareness on the risk of disease | Up to 90 minutes
  Open-ended interviews will be conducted in caregivers of WAS subjects to understand their awareness on the risk of disease (that is, risk of future complications and potential rapid decline).
Number of treatment sequences received by subjects | Up to 90 minutes
  Open-ended interviews will be conducted to understand the treatments received by subjects in terms of sequencing.
Number of subject reported reasons for discontinuation or change in treatment option | Up to 90 minutes
  Open-ended interviews will be conducted in adolescent and adult subjects to understand reasons for discontinuation or change in treatment option for WAS.
Number of caregiver reported reasons for discontinuation or change in treatment option | Up to 90 minutes
  Open-ended interviews will be conducted in caregivers of WAS subjects to understand reasons for discontinuation or change in treatment option for WAS.
Analysis of tolerability of treatment by subjects | Up to 90 minutes
  Open-ended interviews will be conducted in subjects and caregivers to understand the tolerability of WAS treatment by subjects.
Number of subject reported treatment burden | Up to 90 minutes
  Open-ended interviews will be conducted in adolescent and adult subjects to analyze treatment burden for subjects.
Number of caregiver reported treatment burden | Up to 90 minutes
  Open-ended interviews will be conducted in caregivers of WAS subjects to analyze treatment burden for caregivers.
Number of subject reported perspectives on the risk associated with treatment | Up to 90 minutes
  Open-ended interviews will be conducted in adolescent and adult subjects to understand their perspective on the risks associated with each treatment.
Number of caregiver reported perspectives on the risk associated with treatment | Up to 90 minutes
  Open-ended interviews will be conducted in caregivers of WAS subjects to understand their perspective on the risks associated with each treatment.
Number of key concepts of interest | Up to 90 minutes
  Open-ended interviews will be conducted to identify the important concepts of interest that may be used in future clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Collegeville, Pennsylvania, United States

REFERENCES:
- See also: Results for study 208034 can be found on the GSK Clinical Study Register. — https://www.gsk-studyregister.com/study/6052